CLINICAL TRIAL: NCT01130077
Title: A Pilot Study to Evaluate the Effects of Vaccinations with HLA-A2-Restricted Glioma Antigen-Peptides with Poly-ICLC for Children with Newly Diagnosed Malignant Brain Stem Gliomas, Non-Brainstem High-Grade Gliomas, Recurrent Low-Grade Gliomas or Recurrent High Grade Gliomas
Brief Title: A Pilot Study of Glioma Associated Antigen Vaccines in Conjunction with Poly-ICLC in Pediatric Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: James Felker (Other)
Collaborators: Ellie Kavalieros Fund (Unknown); Translational Brain Tumor Research Fund (Unknown); Connor's Cure (Other)
Responsible Party: Sponsor-Investigator, James Felker, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19040319; PRO08030085 (Other: Former identifier from University of Pittsburgh IRB); NCT00862199 (obsolete NCT alias)
Record Dates: First submitted 2010-05-24; First posted 2010-05-25 (Estimated); Last update posted 2024-12-06 (Actual); Status verified 2023-10

CONDITIONS: Newly Diagnosed Pediatric Pontine Glioma; Newly Diagnosed Pediatric High Grade Glioma; Recurrent Pediatric High Grade Glioma; Recurrent Pediatric Low Grade Glioma
Keywords: Pediatric glioma; Vaccine therapy
MeSH Terms: interventions — poly ICLC

STUDY DESIGN:
Intervention Model Description: Pilot study to assess tolerability of this vaccine regimen in different strata of children with high risk gliomas
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HLA Restricted glioma antigen peptides plus Poly ICLC (Experimental): All subjects will receive vaccine plus Poly ICLC will receive 9 injections ( once every 3 weeks)
  Interventions: Biological: HLA-A2 restricted glioma antigen peptides vaccine; Biological: Poly-ICLC

INTERVENTIONS:
Biological: HLA-A2 restricted glioma antigen peptides vaccine — Vaccine given every 3 weeks
  Other Names: BB13624
Biological: Poly-ICLC — Vaccine given every 3 weeks

SUMMARY:
The overall objective of this pilot study is to collect immunological and safety data following administration of vaccinations with HLA-A2. This data will be used to decide whether a larger study of clinical efficacy is warranted.

ELIGIBILITY:
**Inclusion Criteria

*Tumor Types - Tumor type/location:

Stratum A: Newly diagnosed diffuse intrinsic pontine gliomas OR any biopsy proven high-grade glioma* involving the brainstem. Patients may not have received chemotherapy during or after radiation. (Note: Stratum A is closed to accrual.)

Stratum B: Newly diagnosed, non-brainstem high-grade glioma* Patients may not have received chemotherapy during or after radiation. (Note: Stratum B is open to accrual.)

Stratum C: Unresectable low-grade gliomas that have received at least two chemotherapy/biologic regimens. Patients may not have received radiation to the index lesion within 1 year of enrollment. (Note: Stratum C is closed to accrual.)

Stratum D: Non-brainstem high-grade gliomas* that have recurred following treatment. (Note: Stratum D is closed to accrual.)

Stratum E: Newly diagnosed high-grade gliomas* or brain stem gliomas who received chemotherapy during radiation therapy. Patients may not have received chemotherapy after radiation therapy was completed. (Note: Stratum E is closed to accrual.)

Stratum F: Newly diagnosed high-grade gliomas with metastatic disease within the CNS requiring craniospinal radiation therapy. Patients may or may not have received chemotherapy during radiation, but cannot have received chemotherapy after radiation therapy was completed. (Note: Stratum F is closed to accrual.)

* Eligible histologies include glioblastoma (GBM), anaplastic astrocytoma (AA) or gliosarcoma. Patients with any oligodendroglioma component are NOT eligible.
* HLA-A2 positive based on flow cytometry.
* Patients in Stratum A B and E must have received standard involved field radiation therapy [RT] defined as fractionated external beam radiotherapy with total doses between 5000-6000 cGy. Patients in these strata must be registered within 4-12 weeks of completing RT.
* Patients in Stratum F must have received craniospinal radiation.
* Patients must be clinically stable and off or on low-dose (no more than 0.1 mg/kg/day, max 4 mg/day Dexamethasone) corticosteroid for at least one week prior to study registration.
* All patients must sign an IRB-approved informed consent document
* Patients must be ≥ 12 months and <22 years of age at the time of study registration.
* Patients must have a performance status of ≥ to 60.
* Patients must have life expectancy of at least 8 weeks.
* Documented negative serum βHCG for female patients who are post-menarchal. Pregnant females will not be included in the study. Males and females must agree to use effective birth control methods during the course of vaccination.
* Patients must be free of systemic infection.
* Patients with adequate organ function as measured by: Bone marrow: ANC > 1,000/µl; Platelets > 100,000/µl (transfusion independent); absolute lymphocyte count of ≥500/uL; Hemoglobin >8 g/dl (may be transfused). Hepatic: bilirubin ≤ 1.5x institutional normal for age; SGPT (ALT) < 3x institutional normal.

Renal: Serum creatinine based on age or Creatinine clearance or radioisotope GFR >70 ml/min/ml/min/1.73 m²

* Patients on Strata C and D must have recovered from the toxic effects of prior therapy: at least 3 weeks form the last dose of standard cytotoxic chemotherapy or myelosuppressive biological therapy and at least 1 week from the last dose of non-myelosuppressive biologic therapy.
* No overt cardiac, gastrointestinal, pulmonary or psychiatric disease.

Exclusion Criteria:

Patients living outside of North America are not eligible.

Presence of metastatic disease for patients in Stratum A, B, D and E. Patients with low grade gliomas (stratum C) may have tumor spread within the CNS.

Patients in Stratum F must have tumor spread within the CNS.

Patients enrolled in Strata A and B may not have received any prior chemotherapy or anti-glioma therapy of any type other than radiation therapy. Patients enrolled on stratum C must have received at least two prior chemotherapy or biologic therapy regimens and may not have received radiation to the index lesion within 1 year of enrollment. Patients on Strata A, B, E, and F can not have received chemotherapy after radiation therapy was completed.

Concurrent treatment or medications (must be off for at least 1 week) including:

* Interferon (e.g. Intron-A®)
* Allergy desensitization injections
* Growth factors (e.g. Procrit®, Aranesp®, Neulasta®)
* Interleukins (e.g. Proleukin®)
* Any investigational therapeutic medication

Patients must not have a history of, or currently active autoimmune disorders.

Use of immunosuppressives within four weeks prior to study entry. Dexamethasone, or other corticosteroid medications, if used in the peri-operative period and/or during radiotherapy, must be tapered (no more than 0.1 mg/kg/day, max 4 mg/day dexamethasone) for at least one week before study registration. Topical corticosteroids are acceptable.

Patients with known addiction to alcohol or illicit drugs.

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-02; Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Safety: Tolerability during the first two vaccine courses as defined in the protocol. | 6 weeks
  Tolerability during the first two vaccine courses as defined in the protocol.

SECONDARY OUTCOMES:
Glioma-associated antigen-specific T-cell response | Monitoring will continue as long as subject remains on study.
  Glioma-associated antigen-specific T-cell response: determined by IFN-gamma-enzyme linked immune spot (ELISPOT) and tetramer assays

CONTACTS AND LOCATIONS:
Overall Officials: James Felker, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pollack IF, Jakacki RI, Butterfield LH, Hamilton RL, Panigrahy A, Potter DM, Connelly AK, Dibridge SA, Whiteside TL, Okada H. Antigen-specific immune responses and clinical outcome after vaccination with glioma-associated antigen peptides and polyinosinic-polycytidylic acid stabilized by lysine and carboxymethylcellulose in children with newly diagnosed malignant brainstem and nonbrainstem gliomas. J Clin Oncol. 2014 Jul 1;32(19):2050-8. doi: 10.1200/JCO.2013.54.0526. Epub 2014 Jun 2. PMID 24888813
- [Derived] Robison NJ, Kieran MW. Diffuse intrinsic pontine glioma: a reassessment. J Neurooncol. 2014 Aug;119(1):7-15. doi: 10.1007/s11060-014-1448-8. Epub 2014 May 3. PMID 24792486